CLINICAL TRIAL: NCT05259228
Title: Therapeutic Drug Monitoring of Tyrosine Kinase Inhibitor in Patients With Chronic Myeloid Leukemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202008067RIND
Record Dates: First submitted 2022-02-08; First posted 2022-02-28 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Tyrosine Kinase Inhibitor; Pharmacokinetics; Therapeutic Drug Monitoring
Keywords: tyrosine kinase inhibitor; pharmacokinetics; therapeutic drug monitoring

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic myeloid leukemia (CML) consists of 3 clinical stages including chronic phase, accelerated phase and blast crisis. Patients may only survive for few more days to weeks once the disease progresses to blast crisis, even though they might have been stable for several years in the chronic phase. The standard treatment, continuous use of tyrosine kinase inhibitors (TKIs), improves long-term survival, and even may help patients achieve complete remission. Four TKIs are reimbursed by National Health Insurance in Taiwan. Among them, imatinib, nilotinib as well as dasatinib, and ponatinib are the first, second and third generations of TKIs, respectively. Many factors influence the disease control of CML, such as TKI type, genetic mutation and medication adherence. Only 69% of patients followed their physicians' recommendations in a local survey. The medication adherence of TKIs was compromised based on several clinical studies domestically and worldwide due to the slow progression in the chronic phase. Patients might hold or decrease the dose of TKIs on their own when they suffer side effects. Furthermore, the significant intra-subject variations of TKI plasma concentration and drug-drug and drug-food interactions which alter the metabolism of TKIs may lessen therapeutic effect and patient safety. Therefore, this study aims to develop and validate analytic methods of imatinib, dasatinib, nilotinib and ponatinib plasma concentrations. The investigators plan to build the pharmacokinetic models of these 4 TKIs and analyze the impacts of meals, adherence, hepatic enzyme inhibitors and inducers, antacids, proton pump inhibitors and H2 blockers, etc. Adverse drug reactions and treatment outcomes will be evaluated to determine the availability and feasibility of therapeutic drug monitoring of TKIs as part of routine service in pharmacist-led clinics.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥ 20 year-old)
2. Patients who meet the above criteria and have already initiated or are going to receive imatinib, dasatinib, nilotinib, or ponatinib treatment at National Taiwan University Hospital/National Taiwan University Cancer Center from September 2022 to December 2025

Exclusion Criteria:

1. Patients who are unable to cooperate with blood drawing
2. Patients who have not submit the informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥ 20 year-old) who have already initiated or are going to receive imatinib, dasatinib, nilotinib, or ponatinib treatment at National Taiwan University Hospital/National Taiwan University Cancer Center from September 2022 to December 2025.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Analytic methods of TKI plasma concentrations | September, 2022 to December, 2025
  To develop and validate analytic methods of imatinib, dasatinib, nilotinib and ponatinib plasma concentrations.
Minimum plasma concentration [Cmin] of TKI | September, 2022 to December, 2025
  To measure the minimum plasma concentrations of imatinib, dasatinib, nilotinib and ponatinib.
Patient adherence of TKI treatment | September, 2022 to December, 2025
  To follow up and record the adherence of imatinib, dasatinib, nilotinib and ponatinib of each patient.
Analysis of drug-drug interactions | September, 2022 to December, 2025
  To analyze the impacts of hepatic enzyme (CYP) inhibitors and inducers, antacids, proton pump inhibitors and H2 blockers on the concentration of imatinib, dasatinib, nilotinib and ponatinib.
Adverse drug reactions and treatment outcomes of TKI | September, 2022 to December, 2025
  To evaluate the adverse drug reactions and treatment outcomes in order to determine the availability and feasibility of therapeutic drug monitoring of TKIs as part of routine service in pharmacist-led clinics.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Wen Lin, PharmD, MS, Principal Investigator — Graduate Institute of Clinical Pharmacy, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan